CLINICAL TRIAL: NCT02011230
Title: Pain Control as a Function of Hydration Status in the Post Tonsillectomy Patient.
Brief Title: Measuring Pain and Hydration After Tonsillectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB closed study: irregularities in documentation of informed consent, HIPAA
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Angela N Fellner PhD CCRP, Clinical Research Specialist, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13022
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Dehydration
Keywords: Dehydration; Hoist; pain control; The intervention is to provide a commercially available isotonic hydration solution (Hoist®) to the patients.; Patients will drink this solution post procedure as needed.; Patients in the control group will use their discretion to drink any solution they feel suitable
MeSH Terms: conditions — Dehydration; Agnosia | interventions — Lifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients in the control group will not be given any special fluids to take after surgery Patients will use their discretion to drink as needed following surgery
- Hoist (Experimental): Patients in the Hoist group will be given a 10 day supply of Hoist that they will self administer
  Interventions: Other: Hoist Group

INTERVENTIONS:
Other: Hoist Group — Hoist is a commercially available drink that is sold locally. This solution is isotonic meaning that it contains similar concentrations of salt and sugar that are found in the human body
  Other Names: Hoist
  Arms: Hoist

SUMMARY:
Pain after tonsillectomy remains a key barrier during the post operative period. The published return rate to the emergency department for hydration and pain control is approximately 4%. If we can demonstrate decreased pain or decreased visits to the emergency department post tonsillectomy, patient experiences will be improved and health care dollars spent will be decreased. We will attempt to improve hydration status by encouraging consumption of a novel isotonic hydration solution that is currently commercially available.

Our study hypothesis is that patients provided an isotonic hydration solution and instructions on avoiding dehydration post operatively will have improved pain control and decreased emergency department visits.

Improvement in hydration status has the potential of decreasing emergency room visits and subsequent decrease in spending of healthcare dollars. Additional benefits of post-operative hydration may include decrease in pain and decrease in post-operative bleeding rates.

A new isotonic hydration solution with an improved flavor profile (Hoist®) has recently become commercially available. Itis very similar to that of Pedialyte, a commonly used rehydration solution. Pedialyte was designed for rehydration of infants and small children. It has a taste that is not acceptable to many adults and older children.

This study will implement the use of Hoist as suitable rehydration solution. This study is designed to define the relationship between improvement of patient's hydration through provision of a rehydration solution during the post operative period and decrease in complications requiring return to the emergency room, including dehydration and bleeding, as well as improvement in overall pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing tonsillectomy
* Patients undergoing tonsillectomy with adenoidectomy

Exclusion Criteria:

* Patients on anticoagulants
* Patients younger than 3 years old
* Patients with chronic pain syndrome

Ages: 4 Years to 98 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dehydration | 0-10 days
  Patients in the Hoist group will be given a 10 day supply of Hoist (22 bottles). Patients will self-administer the Hoist solution (Parents will administer the Hoist in the case of minor study participants) Pain will be measured during the recovery phase for ten days. Patients will be asked to rate their pain level each day post op (days 0-10) using a numeric pain intensity scale in addition, children ages 4-12 will also receive a Wong-Baker FACES pain scale.

SECONDARY OUTCOMES:
Patient reported pain level | 0-10 days
  Patients will take a survey for up to 10 days after tonsillectomy to rate their level of pain each day. This will be used to see a correlation between reported pain level and amount of fluid intake each day

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schwetschenau, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Queen City ENT, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated